CLINICAL TRIAL: NCT06228183
Title: A Randomized Controlled Trial To Explore the Effect of Intermittent Oro-esophageal Tube Feeding vs. Nasogastric Tube Feeding on Dysphagic Stroke Survivors in Social Interaction and Psychological Status
Brief Title: Effect of Intermittent Oro-esophageal Tube Feeding on Dysphagic Stroke Survivors
Acronym: IOE-xinli
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ethical issues
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024-KY-0115
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experimental group (Experimental): Study lasts 21 days for each patient. The patients were given comprehensive rehabilitation therapy. The experimental group was provided the support of enteral nutrition by Intermittent Oro-esophageal Tube Feeding.
  Interventions: Behavioral: comprehensive rehabilitation therapy; Device: Intermittent Oro-esophageal Tube Feeding
- the control group (Active Comparator): Study lasts 15 days for each patient. The patients were given comprehensive rehabilitation. The control group was provided the support of enteral nutrition by Nasogastric Tube Feeding.
  Interventions: Behavioral: comprehensive rehabilitation therapy; Device: Nasogastric Tube Feeding

INTERVENTIONS:
Behavioral: comprehensive rehabilitation therapy — Both groups were given comprehensive rehabilitation therapy. The main intervention measures included: 1) non-invasive ventilator treatment, generally at least once every night and typically not exceeding continuous daily usage.; 2) attention to feeding and sleeping positions, with a recommended sleeping position of lateral recumbent and the head of the bed raised by 20-30°; 3) swallowing function training, such as tongue muscle stretching training, assisted anterior jaw protrusion training, lemon ice stimulation to the soft palate, pharyngeal wall, etc., generally 5 days per week, twice per day, 5-20 minutes each time; 4) pulmonary ultrashort wave therapy, generally at least 2-3 times a week, and not more than once a day; 5) physical therapy, such as intensive training for gross motor functions including lifting the head, turning over, sitting, crawling, standing, etc., generally 3-5 days per week, 1-2 times per day, 5-20 min each time.
Device: Intermittent Oro-esophageal Tube Feeding — The specific procedure was as follows: the infant was placed in a semi-recumbent or sitting position with the head fixed. Before each feeding, the infant's oral and nasal secretions were to be cleared. An intermittent oro-esophageal tube was appropriately lubricated with water on the head part. The professional medical staff held the tube and slowly inserted it through one side of the mouth into the upper part of the esophagus. The depth of insertion depended on the patient's age and height. After each feeding, the tube was immediately removed, and the patient was held upright for at least 30 minutes in case of reflux.
  Arms: the experimental group
Device: Nasogastric Tube Feeding — Nasogastric Tube Feeding were used for feeding to provide nutritional support. Each feeding was administered by a nurse using the infant's mother's breast milk through the tube. The amount of each feeding varied from 20 to 100 ml depending on the age of the infant, with feedings given every 2 to 3 hours, approximately 10 times per day. The duration of each feeding procedure ranged from 10 to 20 minutes. The total daily intake ranged from 200 to 1000 ml. Each tube was kept indwelling for 5 to 7 days. When the tube needed to be replaced, it was removed after the last feeding of a day and a new tube was to be inserted through the other nostril on the following morning to continue the nutritional support.
  Arms: the control group

SUMMARY:
The goal of this clinical trial is to explore Clinical Effect of Intermittent Oro-esophageal Tube Feeding in Dysphagic Stroke Survivors. The main questions it aims to answer are:

* Can Intermittent Oro-esophageal Tube Feeding improve psychological status in Dysphagic Stroke Survivors?
* Can Intermittent Oro-esophageal Tube Feeding improve social interaction in Dysphagic Stroke Survivors? Patients will be randomly allocated into the control group or the experimental group, all under rehabilitation treatment, the experimental group will be given Intermittent Oro-esophageal Tube Feeding as nutrition support and the control group will be given Nasogastric tube. The study lasts 21 days for each patient. Researchers will compare the Social Functioning Scale, Social Support Questionnaire, Patients Health Questionnaire-9, General Anxiety Disorder-7 to see if the Intermittent Oro-esophageal Tube Feeding can help improve the symptom.

DETAILED DESCRIPTION:
Stroke is happening increasingly more. The goal of this clinical trial is to explore Clinical Effect of Intermittent Oro-esophageal Tube Feeding in Dysphagic Stroke Survivors. The main questions it aims to answer are:

* Can Intermittent Oro-esophageal Tube Feeding improve psychological status in Dysphagic Stroke Survivors?
* Can Intermittent Oro-esophageal Tube Feeding improve social interaction in Dysphagic Stroke Survivors? Patients will be randomly allocated into the control group or the experimental group, all under rehabilitation treatment, the experimental group will be given Intermittent Oro-esophageal Tube Feeding as nutrition support and the control group will be given Nasogastric tube. The study lasts 21 days for each patient. Researchers will compare the Social Functioning Scale, Social Support Questionnaire, Patients Health Questionnaire-9, General Anxiety Disorder-7 to see if the Intermittent Oro-esophageal Tube Feeding can help improve the symptom.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* meeting the diagnostic criteria of stroke;
* any degree of dysphagia at admission;
* steady vital signs, without severe cognitive impairment or sensory aphasia, able to cooperate with the assessment.
* transferred out within three weeks of hospitalization in the neurology department.

Exclusion Criteria:

* complicated with other neurological diseases;
* damaged mucosa or incomplete structure in nasopharynx;
* tracheostomy tube plugged;
* unfeasible to the support of parenteral nutrition;
* simultaneously suffering from liver, kidney failure, tumors, or hematological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Social Functioning Scale | day 1 and day 21
  The Social Functioning Scale includes multiple subscales, and the score range is generally 0-100. Higher scores indicate better social functioning, while lower scores indicate limited social functioning or problems.

SECONDARY OUTCOMES:
Social Support Questionnaire | day 1 and day 21
  Social Support Questionnaire's score range is generally 0-100. Generally, higher scores are better and indicate more social support.
Anxiety | day 1 and day 21
  The anxiety was assessed using the Generalized Anxiety Disorder-7, including items related to fear, worry, attention, etc. The total score ranged from 0 to 21, which was positively correlated with potential anxiety. In the previous study, the scale demonstrated a Cronbach's α-coefficient of 0.879.
Depression | day 1 and day 21
  The depression was assessed using the Patient Health Questionnaire-9, with aspects including mood swings, optimism, sleep quality, appetite, etc. The total score ranged from 0 to 27, which was positively correlated with potential depression. In the previous study, the scale demonstrated a Cronbach's α-coefficient of 0.913.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Zheng da yi fu yuan hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No